CLINICAL TRIAL: NCT06161415
Title: Safety, Tolerability, and Distribution of Topical Laquinimod Eye Drops , an Innovative ImmunomodulatOr Targeting Aryl hydrocarboN Receptor (AhR): The LION Study
Brief Title: Safety, Tolerability, and Distribution of Laquinimod Eye Drops : The LION Study
Acronym: LION
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Quan Dong Nguyen (Other)
Collaborators: Global Ophthalmic Research Center (GORC) (Unknown)
Responsible Party: Sponsor-Investigator, Quan Dong Nguyen, Professor of Ophthalmology, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 71341
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Inflammation; Uveitis
Keywords: Uveitis; Inflammation; Laquinimod eye drops; Topical; Immunomodulation
MeSH Terms: conditions — Inflammation; Uveitis

STUDY DESIGN:
Intervention Model Description: The study will consist of two stages:
  Stage One - Open label dose escalation:
  Up to three subsequent dose-escalation groups will receive Laquinimod eye drops for 2 weeks and samples will be assayed for Laquinimod concentration in aqueous humor, vitreous and plasma.
  Stage Two- Randomized, Controlled Comparison of 2 Laquinimod doses:
  After the dose escalation cohorts are analysed, 2 Laquinimod doses will be selected for a randomized comparison. The doses in stage 2 will not exceed those studied in stage 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): (3 to 6 participants): Participants will receive a dose of Laquinimod as 2 drops once a day (0.6mg per day) in the study eye for 14 days before the surgery.
  Interventions: Drug: Laquinimod eye drops
- Group 2 (Experimental): (3 to 6 participants): Participants will receive a dose of Laquinimod as 2 drops twice a day (1.2mg per day) in the study eye for 14 days before the surgery
  Interventions: Drug: Laquinimod eye drops
- Group 3 (Experimental): (3 to 6 participants): Participants will receive a dose of Laquinimod as 2 drops three times a day(1.8 mg per day) for 14 days before the surgery.
  Interventions: Drug: Laquinimod eye drops
- Stage 2 Comparison Group A (Experimental): (3 to 6 participants): Participants will receive a dose of Laquinimod eye drops in the study eye for 14 days before the surgery. Frequency to be decided at the end of stage 1.
  Interventions: Drug: Laquinimod eye drops
- Stage 2 Comparison Group B (Experimental): (3 to 6 participants): Participants will receive a dose of Laquinimod as 2 drops in the study eye for 14 days before the surgery. Frequency to be decided at the end of stage 1.
  Interventions: Drug: Laquinimod eye drops

INTERVENTIONS:
Drug: Laquinimod eye drops — n Laquinimod eye drops 10 mg/ml Dose: Dosing frequency will depend on the groups assigned
  Other Names: LAQ eye drops

SUMMARY:
The LION Study is a prospective, single-center phase 1 clinical trial to evaluate the safety, tolerability, and distribution of Laquinimod administered as topical eye drops for two weeks in human participants.

DETAILED DESCRIPTION:
Participants who fulfill the study eligibility criteria and who are planned to undergo a pars plana vitrectomy will be enrolled in the study. Eligible participants scheduled for a diagnostic vitrectomy may also be enrolled.

The study will consist of two stages:

Stage One - Open label dose escalation:

Up to three subsequent dose-escalation groups will receive Laquinimod eye drops for 2 weeks and samples will be assayed for Laquinimod concentration in aqueous humor, vitreous and plasma.

Stage Two- Randomized, Controlled Comparison of 2 Laquinimod doses:

After the dose escalation cohorts are analysed, 2 Laquinimod doses will be selected for a randomized comparison. The doses in stage 2 will not exceed those studied in stage 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Participants who are capable and willing to provide informed consent and follow study instructions.
3. Participants who are scheduled to undergo pars plana vitrectomy (PPV).
4. Participants with intraocular pressure (IOP) ≥ 5 mmHg and ≤22 mmHg in study eye
5. Women who are not pregnant or lactating, are post-menopausal or have undergone a sterilization procedure.

Exclusion Criteria:

1. Participants with active periocular or ocular infectious disease (e.g., blepharitis, scleritis, or conjunctivitis, keratitis or endophthalmitis).
2. Participants with active infectious uveitis
3. Participants with a history of prior intraocular or extraocular surgery within 90 days of study enrollment
4. Participant with a history of intravitreal steroids administered to the study eye within 90 days of enrollment.
5. Participants with a history of intravitreal injection of VEGF inhibitors within 30 days of enrollment
6. Use of any topical cyclosporine or corticosteroid or other specified (i.e. calcineurin inhibitors) ophthalmic medication in the study eye for any reason within 14 days of enrollment and before the surgery
7. Use of medication consisting of a strong or moderate inhibitor of CYP3A4 within 2 weeks of Baseline visit (and during the study).
8. Use of medication consisting of a strong inducer of CYP3A4 within 2 weeks of Baseline visit (and during the study)
9. Mild, moderate, or severe hepatic impairment (any of Child-Pugh Score A, B, and C)
10. Moderate or severe renal impairment (GFR ≤60 mL/min)
11. History of HIV disease or other immunodeficiency disorder
12. History of acute hepatitis A (IgM positive), hepatitis B, or hepatitis C
13. History of organ or bone marrow transplant
14. Presence of malignancy under active treatment
15. Any other acute or chronic medical condition that would, in the judgment of the study investigators, reasonably preclude participation in the clinical study
16. Already enrolled in a clinical trial.
17. Any condition that would prevent the investigator from acquiring images of the eye as required per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Concentration of Laquinimod in aqueous humor and vitreous samples of human participants | After 2 weeks of study drug administration
  Assessment of concentration of Laquinimod in aqueous humor and vitreous samples of human by biolanalysis in specialized lab participants on Day 14 of Laquinimod eye-drop administration.
Concentration of Laquinimod in plasma of human participants | After 2 weeks of study drug administration
  Assessment of concentration of Laquinimod in plasma of human participants on Day 14 of Laquinimod in specialized lab eye-drop administration. participants on Day 14 of Laquinimod eye-drop administration.

SECONDARY OUTCOMES:
Safety Assessment | Baseline to end of Study at 22-30days
  Any Adverse events: ocular and non-ocular at Post operative Day 1 and Post operative Day 8 compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Spencer Center for Vision Research at the Byers Eye Institute, Palo Alto, California, United States